CLINICAL TRIAL: NCT05548283
Title: Standardizing Treatments for Pulmonary Exacerbations: A Platform for Evaluating Treatment Decisions to Improve Outcomes (STOP360) Aminoglycoside Study (AG Study)
Brief Title: Standardizing Treatments for Pulmonary Exacerbations - Aminoglycoside Study
Acronym: STOP360AG
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chris Goss (Other)
Collaborators: University of Washington (Other); Medical University of South Carolina (Other); Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor-Investigator, Chris Goss, Associate Director, UW Adult CF Center, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STOP360-IP-22 AG
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis Pulmonary Exacerbation
Keywords: Cystic Fibrosis; CF; Cystic Fibrosis Pulmonary Exacerbation; aminoglycoside; beta-lactam; β-lactam; STOP; STOP360
MeSH Terms: conditions — Cystic Fibrosis | interventions — Monobactams; Aminoglycosides

STUDY DESIGN:
Intervention Model Description: The aminoglycoside study will compare treatment of an IV β-lactam and aminoglycoside (AG) versus an IV β-lactam only (non-AG). Individuals will be randomly assigned in a 1:1 fashion to receive either the AG or non-AG intervention for a planned 14 day course of IV antibiotics. IV antibiotic treatments for each intervention arm will be selected by the treating physician following standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- β-lactam Only (Non-AG) (Other): Participants randomized to this arm will be prescribed a standard of care intravenous (IV) β-lactam as selected by their treating physician. Treatment must not include an IV aminoglycoside.
  Interventions: Drug: Beta-lactam antibiotic
- β-lactam and Aminoglycoside (AG) (Other): Participants randomized to this arm will be prescribed a standard of care intravenous (IV) β-lactam and aminoglycoside selected by their treating physician.
  Interventions: Drug: Beta-lactam antibiotic; Drug: Aminoglycoside

INTERVENTIONS:
Drug: Beta-lactam antibiotic — Intravenous (IV) β-lactam will be selected by the treating physician following standard of care. Treatment will last for 14 days (± 2 days).
  Other Names: β-lactam
Drug: Aminoglycoside — Intravenous (IV) aminoglycoside will be selected by the treating physician following standard of care. Treatment will last for 14 days (± 2 days).
  Other Names: AG
  Arms: β-lactam and Aminoglycoside (AG)

SUMMARY:
The purpose of this study is to look at pulmonary exacerbations in people with cystic fibrosis (CF) that need to be treated with antibiotics given through a tube inserted into a vein (intravenous or IV). A pulmonary exacerbation is a worsening of respiratory symptoms in people with CF that needs medical intervention. Both doctors and CF patients are trying to understand the best way to treat pulmonary exacerbations. This study is trying to answer the following questions about treating a pulmonary exacerbation:

* Do participants have the same improvement in lung function and symptoms if they are treated with one type of antibiotic (called beta-lactams or β-lactams) versus taking two different types of antibiotics (tobramycin and β-lactams)?
* Is taking one type of antibiotic just as good as taking two types?

DETAILED DESCRIPTION:
Cystic Fibrosis Foundation (CFF) treatment guidelines for the management of pulmonary exacerbations (PEx) identified evidence gaps in current clinical best practices. The STOP program offers a platform for the conduct of controlled trials to develop the evidence base in order to define clinical best practices. The interventional Aminoglycoside Study (AG Study) will be a prospective, multi-center, parallel group, randomized (1:1 ratio), open-label, superiority study of intravenous aminoglycoside and β-lactams versus intravenous β-lactams only. Randomization will occur at Visit 1. The primary objective of this platform trial is to evaluate the efficacy and safety of differing treatments in CF PEx during a planned 14 day course of IV antimicrobials. Primary efficacy will be evaluated as the difference in mean Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) changes from Visit 1 to Visit 2 (Day 28 ± 2 days) between intervention arms.

ELIGIBILITY:
Inclusion Criteria:

* All genders ≥ 6 years of age at Visit 1
* Documentation of a CF diagnosis
* Clinician intent to treat index CF PEx with a planned 14-day course of IV antimicrobials
* At least one documented Pa positive culture within two years prior to Visit 1

Exclusion Criteria:

* Participant is not pregnant
* No known renal impairment or history of solid organ transplantation
* No IV antimicrobial treatment, ICU admission, pneumothorax, or hemoptysis within 6 weeks prior to Visit 1
* No use of investigational therapies, new CF transmembrane conductance regulator (CFTR) modulators, or treatment for Nontuberculous mycobacteria (NTM) within 4 weeks prior to Visit 1
* No history of hypersensitivity, vestibular, or auditory toxicity with aminoglycosides
* No more than one day of IV aminoglycosides administered for the current PEx treatment prior to Visit 1

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 730 (Estimated)
Dates: Start 2023-04-23 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Absolute Change in FEV1 % Predicted at Week 4 in Aminoglycoside (AG) Study | Four weeks
  Difference between aminoglycoside (AG) study intervention arms (AG - Non-AG) in the absolute change in FEV1 % predicted from Week 0 (Day 0) to Week 4 (Day 28 ± 2 days)
Incidence of Adverse Events (AEs) in Aminoglycoside (AG) Study Intervention Arms | Six Weeks
  Difference between aminoglycoside (AG) study intervention arms (AG - Non-AG) in the proportion of participants with at least one AE from Week 0 (Day 0) to Week 6 (Day 44 ± 2 days).

SECONDARY OUTCOMES:
Absolute Change in CFRSD-CRISS Score at Week 4 in Aminoglycoside (AG) Study | Four weeks
  Difference between aminoglycoside (AG) study intervention arms (AG - Non-AG) in the absolute change in respiratory symptoms, as measured by the CF Respiratory Symptoms Diary-Chronic Respiratory Infection Symptom Score (CFRSD-CRISS) from Week 0 (Day 0) to Week 4 (Day 28 ± 2 days). The CFRSD-CRISS is derived from a set of questions asking a participant to state the extent of their 8 respiratory symptoms: difficulty breathing, feverishness, tiredness, chills or sweats, coughing, coughing up mucus, tightness in the chest and wheezing. Each respiratory symptom is assigned a score from 0-4 based on the response, with zero corresponding to the absence of the symptom and four corresponding to symptom being present 'a great deal' or 'extremely'. A summed score (range from 0-24) is calculated for each participant and converted to a final score with a range of 0 to 100, where the lowest scores indicate improvement of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Flume, MD, Principal Investigator — Medical University of South Carolina
Locations (60):
- United States (59):
  - The Children's Hospital Alabama, University of Alabama at Birmingham, Birmingham, Alabama
  - Tucson Cystic Fibrosis Center, Tucson, Arizona
  - University of California San Diego, La Jolla, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - CHOC Children's Hospital, Orange, California
  - University of California at Davis Medical Center, Sacramento, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Emory University, Atlanta, Georgia
  - Saint Luke's Cystic Fibrosis Center of Idaho, Boise, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Maine Medical Center, Portland, Maine
  - John Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Brigham & Women's Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - University of Michigan, Michigan Medicine, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - SSM Health Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Lenox Hill Hospital Cystic Fibrosis Center, New York, New York
  - Children's Hospital of New York, New York, New York
  - New York Medical College at Westchester Medical Center, Valhalla, New York
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - Oklahoma Cystic Fibrosis Center, Oklahoma City, Oklahoma
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - University of Texas Southwestern / Children's Health, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Providence Medical Group, Cystic Fibrosis Clinic, Spokane, Washington
  - West Virginia University - Morgantown, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
- University of Calgary Adult Cystic Fibrosis Clinic (Calgary, AB), Calgary, Alberta, Canada